CLINICAL TRIAL: NCT00126022
Title: A Multi-Center, Double-Blind, Randomized, Placebo-Controlled, Parallel Design Study to Evaluate the Efficacy and Safety of Intravenous Tedisamil Sesquifumarate in the Rapid Conversion to Normal Sinus Rhythm in Female Subjects With Recent Onset Atrial Fibrillation
Brief Title: Intravenous Tedisamil in the Rapid Conversion of Atrial Fibrillation or Flutter to Normal Sinus Rhythm in Female Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S219.3.116; 2004-000460-27
Record Dates: First submitted 2005-08-01; First posted 2005-08-02 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2006-03

CONDITIONS: Atrial Fibrillation; Atrial Flutter
Keywords: Atrial fibrillation; atrial flutter; anti-arrhythmic agents; conversion to normal sinus rhythm
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter

INTERVENTIONS:
Drug: Tedisamil sesquifumarate

SUMMARY:
The purpose of this study is to demonstrate the ability of tedisamil to convert atrial fibrillation or flutter into normal sinus rhythm (NSR) in female patients.

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign informed consent before screening examinations are performed and before the study drug is administered
* Females > 18 years of age
* Subjects with documented (60 second rhythm strip) symptomatic atrial fibrillation or flutter (duration > 3 hours and < 45 days) at the time of randomization
* Subjects who are in no distress and hemodynamically stable (supine systolic blood pressure > 90 mmHg and diastolic blood pressure < 105 mmHg)

Exclusion Criteria:

* Pregnancy and lactation
* Acute myocardial infarction and cerebrovascular accidents
* Coronary syndromes and congestive heart failure (CHF) New York Heart Association (NYHA) IV
* Life-threatening ventricular arrhythmias and electrocardiogram (ECG) abnormalities
* Concurrent antiarrhythmic treatments

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-12; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (81):
- Site 82, Tullahoma, Tennessee, United States
- Argentina (4):
  - Site 2, Buenos Aires
  - Site 3, Buenos Aires
  - Site 5, Munro
  - Site 4, San Miguel de Tucumán
- Czechia (9):
  - Site 8, Brno
  - Site 11, Jindřichův Hradec
  - Site 9, Ostrava-Poruba
  - Site 10, Pilsen
  - Site 14, Prague
  - Site 6, Prague
  - Site 7, Prague
  - Site 12, Slaný
  - Site 13, Ústí nad Orlicí
- Germany (3):
  - Site 15, Bad Nauheim
  - Site 17, Göttingen
  - Site 16, Halle
- Israel (6):
  - Site 18, Haifa
  - Site 19, Jerusalem
  - Site 22, Jerusalem
  - Site 23, Jerusalem
  - Site 20, Tel Aviv
  - Site 21, Tel Aviv
- Poland (13):
  - Site 26, Bydgoszcz
  - Site 32, Bydgoszcz
  - Site 30, Lodz
  - Site 29, Lublin
  - Site 36, Lublin
  - Site 31, Medyczna
  - Site 33, Szczecin
  - Site 24, Warsaw
  - Site 25, Warsaw
  - Site 27, Warsaw
  - Site 28, Warsaw
  - Site 34, Wroclaw
  - Site 35, Wroclaw
- Romania (4):
  - Site 38, Brasov
  - Site 39, Bucharest
  - Site 40, Bucharest
  - Site 37, Tg. Mures
- Russia (11):
  - Site 41, Moscow
  - Site 42, Moscow
  - Site 43, Moscow
  - Site 44, Moscow
  - Site 45, Moscow
  - Site 46, Moscow
  - Site 47, Moscow
  - Site 48, Moscow
  - Site 49, Moscow
  - Site 51, Moscow
  - Site 50, Saint Petersburg
- Serbia and Montenegro (7):
  - Site 52, Belgrade
  - Site 53, Belgrade
  - Site 54, Belgrade
  - Site 57, Belgrade
  - Site 58, Belgrade
  - Site 56, Niska Banja
  - Site 55, Sremska Kamenica
- Slovakia (7):
  - Site 60, Banská Bystrica
  - Site 64, Bratislava
  - Site 61, Košice
  - Site 62, Lučenec
  - Site 59, Nitra
  - Site 65, Nové Zámky
  - Site 63, Prešov
- South Africa (2):
  - Site 66, Cape Town
  - Site 67, Cape Town
- Ukraine (13):
  - Site 68, Dnipro
  - Site 69, Dnipro
  - Site 71, Donetsk
  - Site 72, Donetsk
  - Site 75, Kharkiv
  - Site 70, Kiev
  - Site 73, Kiev
  - Site 76, Kiev
  - Site 77, Kiev
  - Site 74, Lviv
  - Site 80, Odesa
  - Site 79, Zaporizhya
  - Site 78, Zaporizhzhya
- Site 81, London, United Kingdom